CLINICAL TRIAL: NCT06651411
Title: The Feasibility of Chatbot-based Stress Management Intervention STARS for Youth in Lithuania: a Pilot Randomized Controlled Trial
Brief Title: The Feasibility of Chatbot-based Stress Management Intervention STARS for Youth in Lithuania
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vilnius University (Other)
Collaborators: World Health Organization (Other)
Responsible Party: Principal Investigator, Evaldas Kazlauskas, Professor in clinical psychology, Vilnius University
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: (1.13E)250000-KT-67/ERC0004137
Record Dates: First submitted 2024-10-17; First posted 2024-10-21 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2024-10

CONDITIONS: Symptoms of Depression and Anxiety
Keywords: Intervention; Chatbot; Stress management; youth; STARS; Feasibility
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): The intervention group will get a 10-session chatbot-based stress management intervention.
  Interventions: Behavioral: STARS (Scalable Technology for Adolescents and youth to Reduce Stress)
- Control group (Other): The control group will get basic psychoeducation.
  Interventions: Behavioral: Basic psychoeducation

INTERVENTIONS:
Behavioral: STARS (Scalable Technology for Adolescents and youth to Reduce Stress) — The intervention is a chatbot-based stress management intervention developed by the World Health Organization (WHO). It consists of 10 sessions, which include: Introduction (1), Psychoeducation (2), Emotion Regulation (3, 4), Behavior Activation (5, 6), Managing Problems (7), Thought Challenging (8, 9), and Relapse Prevention (10). Each session consists of psychoeducation and exercise parts. Trained e-helpers contact participants to support them individually weekly.
  The effect of the intervention will be compared against a control group that receives basic psychoeducation. The intervention is provided in Lithuanian.
  Arms: Intervention group
Behavioral: Basic psychoeducation — Basic psychoeducation includes basic information on stress management.
  Arms: Control group

SUMMARY:
The study aims to assess the feasibility of a chatbot-based stress management intervention among youth in Lithuania.

DETAILED DESCRIPTION:
The intervention is a chatbot-based stress management intervention developed by the World Health Organization (WHO). It consists of 10 sessions which include: Introduction (1), Psychoeducation (2), Emotion Regulation (3, 4), Behavior Activation (5, 6), Managing Problems (7), Thought Challenging (8, 9), and Relapse Prevention (10). Each session consists of psychoeducation and exercise parts. Trained e-helpers contact participants to support them individually on a weekly basis.

The effect of the intervention will be compared against a control group which gets basic psychoeducation. The intervention is provided in Lithuanian.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18-25 years
* Understanding the Lithuanian language
* Having access to a device for intervention delivery
* Experiencing moderate levels of psychological distress

Exclusion Criteria:

* People at imminent risk of suicide
* People currently experiencing a psychotic episode
* People currently experiencing interpersonal violence
* Current dependency on alcohol/drugs

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2024-10-30 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Changes in The Patient Health Questionnaire-9 | Before the intervention, immediately after the intervention, 3-months after the intervention
  Changes in symptoms of depression are measured. The Patient Health Questionnaire-9 (PHQ-9, Kroenke et al., 2001) is a self-report measure comprising 9 items about symptoms of depression. All items are answered on a 4-point Likert scale that ranges from 0 (not at all) to 3 (nearly every day). A higher score indicates more pronounced symptoms.
Changes in The Generalized Anxiety Disorder-7 | Before the intervention, immediately after the intervention, 3-months after the intervention
  Changes in symptoms of anxiety are measured. The Generalized Anxiety Disorder-7 (GAD-7, Spitzer et al., 2006) is a self-report measure comprising 7 items about symptoms of anxiety. All items are answered on a 4-point Likert scale that ranges from 0 (not at all) to 3 (nearly every day). A higher score indicates more pronounced symptoms.

SECONDARY OUTCOMES:
Changes in Kessler-6 | Before the intervention, immediately after the intervention, 3-months after the intervention
  Changes in psychological distress are measured. Kessler-6 (K6, Kessler et al., 2002) is a self-report measure comprising 6 questions about psychological distress. All items are answered on a 5-point Likert scale that ranges from 0 (none of the time) to 4 (all of the time). A higher score indicates more pronounced symptoms.
Changes in The Brief Adjustment Disorder Measure-8 | Before the intervention, immediately after the intervention, 3-months after the intervention
  Changes in symptoms of adjustment disorder are measured. The Brief Adjustment Disorder Measure-8 (ADNM-8, Kazlauskas et al., 2018) is a self-report measure comprising 8 items about symptoms of adjustment disorder. All items are answered on a 4-point Likert scale that ranges from 1 (never) to 4 (often). A higher score indicates more pronounced symptoms.
Changes in The SIDAS | Before the intervention, immediately after the intervention, 3-months after the intervention
  Changes in suicidal ideation are measured. The SIDAS (Van Spijker et al., 2014) is a self-report measure comprising 5 questions about suicidal ideation. All items are answered on a 10-point Likert scale that ranges from 0 (never, no control, not close at all, not at all) to 10 (always, full control, made an attempt, extremely). A higher score indicates more pronounced symptoms.
Changes in The WHODAS 2.0 | Before the intervention, immediately after the intervention, 3-months after the intervention
  Changes in functioning are measured. The WHODAS 2.0 (Ustun et al., 2010) is a self-report measure comprising 12 questions about functioning. All items are answered on a 5-point Likert scale that ranges from 0 (none) to 4 (extreme or cannot do). A higher score indicates more pronounced symptoms.
Changes in The World Health Organization Well-being Index-5 | Before the intervention, immediately after the intervention, 3-months after the intervention
  Changes in psychological well-being are measured. The World Health Organization Well-being Index-5 (WHO-5, Bech, 2004) is a self-report measure comprising 5 items about psychological well-being. All items are answered on a 5-point Likert scale that ranges from 0 (at no time) to 4 (all of the time). A higher score indicates more pronounced psychological well-being.
Changes in The International Trauma Questionnaire | Before the intervention, immediately after the intervention, 3-months after the intervention
  Changes in symptoms of post-traumatic stress disorders are measured. International Trauma Questionnaire (ITQ, Cloitre et al., 2018) is a self-report measure comprising 18 items. All items are answered on a 5-point Likert scale that ranges from 0 (not at all) to 4 (extremely). A higher score indicates more pronounced symptoms.
Changes in The Resilience scale | Before the intervention, immediately after the intervention, 3-months after the intervention
  Changes in resilience are measured. The Resilience scale (RS-14, Wagnild, 2011) is a self-report measure comprising 14 items about resilience. All items are answered on a 7-point Likert scale that ranges from 1 (strongly disagree) to 7 (strongly agree). A higher score indicates more pronounced resilience.
Changes in The Client Services Receipt Inventory | Before the intervention, 3-months after the intervention
  Changes in client service are measured. The Client Services Receipt Inventory (CSRI, Beeacham and Knapp, 2001) is a self-report measure comprising questions about client service. The CSRI covers a broad range of services that may be utilized, including primary and secondary care services, other services, and informal care.
Changes in The EQ-5D-5L | Before the intervention, immediately after the intervention, 3-months after the intervention
  Changes in health are measured. The EQ-5D-5L (EuroQol Research Foundation, 2019) is a self-report measure comprising 5 items about health. All items are answered on a 5-point Likert scale that ranges from 1 (I have no problems or similar) to 5 (I am unable or similar). A higher score indicates more pronounced symptoms.
Recruitment rate | Before the intervention
  Recruitment rate recorded as the number of eligible participants who consent to participate in the study will be assessed.
Drop-out rates | Immediately after the intervention, 3-months after the intervention
  Drop-out rates recorded as the number of randomized participants who do not complete the intervention, the post-test assessment, and three-month follow-up assessment will be assessed.
Number of adverse events and serious adverse events | Immediately after the intervention
  Number of adverse events and serious adverse events will be assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- Vilnius University, Vilnius, Lithuania

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data can be shared upon a reasonable request.